CLINICAL TRIAL: NCT00305487
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Clinical Trial Designed to Assess the Safety and Efficacy of Ciclesonide (200mcg and 100mcg, Once Daily) Applied as a Nasal Spray for Two Weeks in the Treatment of Seasonal Allergic Rhinitis (SAR) in Patients 6 to 11 Years of Age
Brief Title: Safety and Efficacy of Ciclesonide in Pediatric Patients (6 to 11 Years of Age) With Seasonal Allergic Rhinitis (BY9010/M1-417)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-417
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Hay Fever; Seasonal Allergic Rhinitis
Keywords: Hay Fever; Seasonal Allergic Rhinitis; Nasal spray; Ciclesonide; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

INTERVENTIONS:
Drug: Ciclesonide nasal spray

SUMMARY:
The aim of the study is to determine the efficacy and safety of ciclesonide nasal spray in children with seasonal allergic rhinitis. Ciclesonide will be administered intranasally at two dose levels once daily. The study consists of a baseline period (1 to 3 weeks) and a treatment period (2 weeks).

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* General good health other than seasonal allergic rhinitis
* Positive standard skin prick test

Main Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes for in vitro fertilization
* Participation in any investigational drug trial within the 30 days preceding the Screening Visit
* A known hypersensitivity to any corticosteroid or any of the ingredients in the study drug formulation
* Plans to travel outside the study area (the known pollen area for the investigative site) for 24 hours or more during the final 7 days of the baseline period
* Plans to travel outside the study area (the known pollen area for the investigative site) for more than 2 consecutive days OR more than 3 days total during the treatment period
* Use of any prohibited concomitant medications
* Non-vaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding the Screening Visit
* Use of antiepileptic drugs for epilepsy within 30 days of the Screening Visit
* Study participation by more than one patient from the same household

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 660
Dates: Start 2006-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Average of morning and evening parent/caregiver reported reflective total nasal symptoms score over the two weeks of treatment

SECONDARY OUTCOMES:
Physician assessment of nasal symptoms score at endpoint
average of morning and evening parent/caregiver reported instantaneous total nasal symptom score over the two weeks of treatment
safety

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (68):
- United States (68):
  - Altana Pharma/Nycomed, Birmingham, Alabama
  - Altana Pharma/Nycomed, Hot Springs, Arkansas
  - Altana Pharma/Nycomed, Costa Mesa, California
  - Altana Pharma/Nycomed, Huntington Beach, California
  - Altana Pharma/Nycomed, Long Beach, California
  - Altana Pharma/Nycomed, Los Alamitos, California
  - Altana Pharma/Nycomed, Mission Viejo, California
  - Altana Pharma/Nycomed, Orange, California
  - Altana Pharma/Nycomed, Roseville, California
  - Altana Pharma/Nycomed, San Diego, California
  - Altana Pharma/Nycomed, San Jose, California
  - Altana Pharma/Nycomed, Stockton, California
  - Altana Pharma/Nycomed, Colorado Springs, Colorado
  - Altana Pharma/Nycomed, Denver, Colorado
  - Altana Pharma/Nycomed, Englewood, Colorado
  - Altana Pharma/Nycomed, Lakewood, CO, Colorado
  - Altana Pharma/Nycomed, Atlanta, Georgia
  - Altana Pharma/Nycomed, Gainesville, Georgia
  - Altana Pharma/Nycomed, Savannah, Georgia
  - Altana Pharma/Nycomed, Woodstock, GA, Georgia
  - Altana Pharma/Nycomed, Normal, Illinois
  - Altana Pharma/Nycomed, Indianapolis, Indiana
  - Altana Pharma/Nycomed, Overland Park, Kansas
  - Altana Pharma/Nycomed, Louisville, KY, Kentucky
  - Altana Pharma/Nycomed, Metairie, Louisiana
  - Altana Pharma/Nycomed, Shreveport, Louisiana
  - Altana Pharma/Nycomed, Bethesda, Maryland
  - Altana Pharma/Nycomed, North Dartmouth, Massachusetts
  - Altana Pharma/Nycomed, Minneapolis, Minnesota
  - Altana Pharma/Nycomed, Jefferson City, Missouri
  - Altana Pharma/Nycomed, Rolla, Missouri
  - Altana Pharma/Nycomed, St Louis, Missouri
  - Altana Pharma/Nycomed, Lincoln, NE, Nebraska
  - Altana Pharma/Nycomed, Papillion, Nebraska
  - Altana Pharma/Nycomed, Brick, New Jersey
  - Altana Pharma/Nycomed, Forked River, New Jersey
  - Altana Pharma/Nycomed, Red Bank, New Jersey
  - Altana Pharma/Nycomed, Skillman, New Jersey
  - Altana Pharma/Nycomed, Warren Township, New Jersey
  - Altana Pharma/Nycomed, Rochester, NY, New York
  - Altana Pharma/Nycomed, Rockville Centre, New York
  - Altana Pharma/Nycomed, Raleigh, North Carolina
  - Altana Pharma/Nycomed, Cincinnati, Ohio
  - Altana Pharma/Nycomed, Cincinnati, OH, Ohio
  - Altana Pharma/Nycomed, Ashland, Oregon
  - Altana Pharma/Nycomed, Lake Oswego, Oregon
  - Altana Pharma/Nycomed, Medford, OR, Oregon
  - Altana Pharma/Nycomed, Portland, Oregon
  - Altana Pharma/Nycomed, Blue Bell, Pennsylvania
  - Altana Pharma/Nycomed, Eerie, Pennsylvania
  - Altana Pharma/Nycomed, Pittsburgh, Pennsylvania
  - Altana Pharma/Nycomed, Upland, Pennsylvania
  - Altana Pharma/Nycomed, Charleston, South Carolina
  - Altana Pharma/Nycomed, Charleston, SC, South Carolina
  - Altana Pharma/Nycomed, Germantown, Tennessee
  - Altana Pharma/Nycomed, Jackson, Tennessee
  - Altana Pharma/Nycomed, Austin, Texas
  - Altana Pharma/Nycomed, Dallas, Texas
  - Altana Pharma/Nycomed, El Paso, Texas
  - Altana Pharma/Nycomed, Kerrville, Texas
  - Altana Pharma/Nycomed, New Braunfels, Texas
  - Altana Pharma/Nycomed, San Antonio, Texas
  - Altana Pharma/Nycomed, Salt Lake City, Utah
  - Altana Pharma/Nycomed, South Burlington, Vermont
  - Altana Pharma/Nycomed, Burke, Virginia
  - Altana Pharma/Nycomed, Charlottesville, Virginia
  - Altana Pharma/Nycomed, Richmond, Virginia
  - Altana Pharma/Nycomed, Milwaukee, Wisconsin

REFERENCES:
- See also: BY9010-M1-417-RDS-2007-04-27.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4540&filename=BY9010-M1-417-RDS-2007-04-27.pdf